CLINICAL TRIAL: NCT03596983
Title: P20 Extending Sleep to Reverse Metabolic Syndrome in Middle-Aged Adults: Acceptability and Feasibility of a Sleep Intervention
Brief Title: P20 Extending Sleep to Reverse Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-00707
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome
Keywords: sleep intervention; metabolic syndrome; hypertension; type 2 diabetes; abdominal obesity; dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Diabetes Mellitus, Type 2; Obesity, Abdominal; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short Sleep Patients (Experimental): Intervention: Self-management for Adequate Sleep Intervention (SASI). SASI was developed Dr. Michael Grandner. SASI is based on Cognitive Behavioral Therapy for Insomnia (CBTI), an established and effective approach for treating insomnia. Like CBTI, SASI extends sleep duration based on sleep efficiency (the proportion of time spent sleeping during a sleep episode). Bed times and wake times will be prescribed each week for each participant and allow for gradual increases in sleep opportunity. Bedtimes will be set 15 minutes earlier each week provided sleep efficiency remains >90%. Earlier betimes will extend sleep duration by increasing the opportunity for sleep. Wake times will not be changed because wake times are often determined by external demands, such as work schedules.
  Interventions: Behavioral: Sleep Intervention; Behavioral: Week 2 Intervention

INTERVENTIONS:
Behavioral: Sleep Intervention — * Sleep Diaries (Daily)
  * Fitbit 24/7
  * Phone/ video conference calls (weekly with study team)
  * Epworth Sleepiness Scale (weekly)
  * PROMIS fatigue scale-evening (weekly)
Behavioral: Week 2 Intervention — * Sleep Diaries (Daily)
  * Phone Calls (weekly with study team)
  * Wrist Accelerometry and fitbit 24/7 for 14 days
  * SAFTEE Questionnaire
  * ASA24
  * Behavioral risk factor surveillance system (smoking and alcohol use questions)
  * Psychological well-being (SF36)
  * Index of Self Regulation
  * PROMIS fatigue scale-morning (weekly)
  * PROMIS fatigue scale-evening (weekly)
  * Epworth Sleepiness Scale (weekly)

SUMMARY:
This pilot study will test the acceptability and feasibility of a sleep extension intervention in community-dwelling, short-sleeping, racially/ethnically diverse middle-aged adults with MetS. Baseline sleep habits will be assessed and used to guide individualized strategies to extend sleep. A 1-group pretest-posttest study design will test the efficacy of this 18-week study (2 weeks of baseline data collection, 1 week of study intervention planning, 12 weeks of sleep intervention delivery, final follow up 3 weeks after last day of the 12-week intervention) on sleep duration, MetS risk behaviors (reduced physical activity, increased sedentary behavior, poor diet quality), symptoms associated with MetS risk behaviors (poor affective well-being, fatigue), and self-regulation. Socio-ecological barriers and facilitators to the intervention will be identified using a quantitative and qualitative approac

DETAILED DESCRIPTION:
Screening and consent process. Potential participants will be informed about the study, provide verbal consent to be screened, and begin a multi-stage screening process consisting of a screening questionnaire (in person or by phone), an intake visit, and a home sleep test (OSA, sleep duration). The screening questionnaire will assess inclusion/exclusion criteria including demographics (NINR Demographic data), sleep duration and timing (STQ)70, insomnia symptoms (ISI), OSA symptoms (MAP), depressive symptoms (PROMIS depression v1.0), alcohol abuse (AUDIT), and self-reported habitual napping, sleep-promoting medication use, recent or planned shift work or trans-meridian travel, pregnancy/lactation, and current chemotherapy. Individuals meeting inclusion criteria based on the screening questionnaire will be invited to the CTSI visit. During the CTSI visit, the study team will describe the study and obtain written informed consent. MetS diagnosis will be confirmed based on measures of waist circumference, fasting glucose, serum triglycerides, high density lipoprotein cholesterol (HDL-c), and resting blood pressure. Waist circumference will assessed as the mean of 3 measurements taken at the level of the umbilicus using non-distensible measuring tape. Blood pressure will be assessed as the average of 3 recordings each taken 1 minute apart, following 10 minutes of inactivity. A 4th recording will occur if any two systolic or diastolic readings are >5 mmHg apart. Fasting glucose, serum triglycerides, and HDL-c will be measured from blood samples drawn according to standard venipuncture protocol at the CTSI. Analysis will be completed at the CTSI lab using standard techniques for analyzing the blood samples. Retained participants will be trained to use a home sleep apnea testing device (Embletta MPR) to objectively screen for OSA, a wrist accelerometer, and a sleep diary to screen for short sleep. Written instructions and study team contact information will be provided. Participants will return the home sleep apnea testing device in a prepaid package. Data will be downloaded from the home sleep apnea testing device and scored by a sleep technician to confirm the absence of moderate/severe OSA (AHI ≥15).

Baseline data collection. Retained participants will complete the remaining baseline measures for sleep duration, MetS risk behaviors (physical activity, sedentary behavior, diet quality, smoking, and alcohol use), sleep deprivation symptoms (quality of life/affective well-being, fatigue) and self-regulation. After baseline week 2, the study team will contact participants to remind them to return the accelerometer in the prepaid shipping package. Participants meeting all the inclusion criteria will be invited to participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 35 years of age and less than or equal to 60 years of age. Middle aged adults have the highest prevalence of short sleep compared to other stages of adulthood.
* Objectively confirmed MetS defined by three or more of the following: a) waist circumference greater than 120cm (men) or 88cm (women), b) blood pressure greater than or equal to 135 mmHg systolic or greater than or equal to 85 mmHg diastolic or antihypertensive medication use, c) fasting glucose greater than or equal to 110 mg/dL or insulin or oral hypoglycemic medication use, d) serum triglycerides greater than or equal to 150mg/dL or hypertriglyceride medication use, e) HDL-c less than 40mg/dL (women) or less than 50 mg/dL (men) or medication use for low HDL-c1. MetS was selected because individuals with MetS are at high risk for multiple chronic conditions.
* Accelerometry confirmed short sleep (average work day sleep less than or equal to 6.5 hours/night). Self-reported sleep may overestimate sleep duration. This will ensure that participants will have short sleep patterns that are associated with MetS outcomes.
* English speaking. Participants will need to demonstrate adequate English comprehension (assessed during informed consent).

Exclusion Criteria:

* Pregnancy/lactation (self-reported). Pregnancy and lactation can disrupt habitual sleep patterns, and hormonal changes during pregnancy increase insulin resistance and may confound MetS.
* Current chemotherapy treatments (self-reported). Current chemotherapy treatments may contribute to fatigue and sleep disturbances.
* Alcohol abuse/dependence will be assessed with the Alcohol Use Disorders Identification Test (a measure that has demonstrated good reliability and validity). Alcohol abuse/dependence may contribute to sleep disturbances and limit the participant's ability to take part in sleep interventions.
* Night shift or shift work (previous 2 months), trans-meridian travel (previous 4 weeks), or planned shift work or trans-meridian travel during intervention period (self-reported). These will be to ensure that sleep estimates from baseline represent participants' habitual sleep and to ensure adherence with the sleep intervention.
* Moderate-severe or severe depression will be assessed with the PHQ-9. Moderate-severe depression or severe depression may contribute to sleep disturbances and interfere with the participant's ability to adhere to the sleep interventions.
* Chronic use of sleep-promoting medications (self-reported). These may interfere with sleep patterns and limit the participant's ability to take part in the sleep interventions.
* Habitual napping, defined as 2 naps per day or > 90 minutes of napping on 3 or more days of the week will be assessed during baseline with accelerometry. This will be to ensure adherence with the sleep intervention.
* Diagnosed but untreated obstructive sleep apnea.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Malone, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after all publications and presentations of the aims for this study are completed.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Malone SK, Patterson F, Grunin L, Goyal C, Hu J, Perez NB, Munroe K, Dickson VV, Melkus GD. Single-arm pilot study of racial differences in sleep extension intervention outcomes among middle-aged adults at risk for metabolic syndrome. J Behav Med. 2026 Jan 13. doi: 10.1007/s10865-025-00624-4. Online ahead of print. PMID 41528656
- [Derived] Malone SK, Patterson F, Hu J, Goyal C, Goel N, Vaughan Dickson V, D'Eramo Melkus G, Aouizerat B. Association between dim light melatonin onset predicted from gene expression profiles with sleep time and chronotype preference: A pilot study. Chronobiol Int. 2025 Oct;42(10):1350-1359. doi: 10.1080/07420528.2025.2546006. Epub 2025 Aug 22. PMID 40844144
- [Derived] Wright F, Malone SK, Wong A, D'Eramo Melkus G, Dickson VV. Addressing Challenges in Recruiting Diverse Populations for Research: Practical Experience From a P20 Center. Nurs Res. 2022 May-Jun 01;71(3):218-226. doi: 10.1097/NNR.0000000000000577. Epub 2022 Jan 24. PMID 35067645

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Sleep Patients: Intervention: Self-management for Adequate Sleep Intervention (SASI). SASI was developed Dr. Michael Grandner. SASI is based on Cognitive Behavioral Therapy for Insomnia (CBTI), an established and effective approach for treating insomnia. Like CBTI, SASI extends sleep duration based on sleep efficiency (the proportion of time spent sleeping during a sleep episode). Bed times and wake times will be prescribed each week for each participant and allow for gradual increases in sleep opportunity. Bedtimes will be set 15 minutes earlier each week provided sleep efficiency remains >90%. Earlier betimes will extend sleep duration by increasing the opportunity for sleep. Wake times will not be changed because wake times are often determined by external demands, such as work schedules.
  Sleep Intervention: - Sleep Diaries (Daily)
  * Fitbit 24/7
  * Phone/ video conference calls (weekly with study team)
  * Epworth Sleepiness Scale (weekly)
  * PROMIS fatigue scale-evening (weekly)
  Week 2 Intervention: - Sleep Diaries (Daily)
  * Phone Calls (weekly with study team)
  * Wrist Accelerometry and fitbit 24/7 for 14 days
  * SAFTEE Questionnaire
  * ASA24
  * Behavioral risk factor surveillance system (smoking and alcohol use questions)
  * Psychological well-being (SF36)
  * Index of Self Regulation
  * PROMIS fatigue scale-morning (weekly)
  * PROMIS fatigue scale-evening (weekly)
  * Epworth Sleepiness Scale (weekly)
Period: Overall Study
Arm/Group | Short Sleep Patients
Started | 44
Completed | 41
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 21
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: SASI Acceptability Questionnaire Score at Pre-Intervention
Description: 14-item questionnaire assessing acceptability of SASI. Items are ranked on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score is the average item score and ranges from 1-5. Higher total scores indicate greater overall acceptability.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 44
score on a scale | 3.91 (0.37)

2. Primary Outcome: SASI Acceptability Questionnaire Score at Post-Intervention
Description: as for outcome 1
Time Frame: Week 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
score on a scale | 4.3 (0.37)

3. Primary Outcome: Recruitment Rate
Description: The percentage of screened participants who were enrolled in the study.
Time Frame: Baseline
Measure: Number; unit: Percentage of participants
Groups:
- Screened Participants: Participants who were screened for enrollment in the study.
Arm/Group | Screened Participants
Number analyzed (Participants) | 81
Percentage of participants | 54

4. Primary Outcome: Retention Rate
Description: Percentage of Enrolled Participants who completed the 15-Week intervention.
Time Frame: Up to Week 15
Measure: Number; unit: Percentage of participants
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 44
Percentage of participants | 93

5. Primary Outcome: Protocol Adherence Rate
Description: The percentage of participants completing greater than or equal to 4 daily sleep diary entries per week for 80% or more of the intervention period.
Time Frame: Week 15
Measure: Number; unit: Percentage of participants
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
Percentage of participants | 99

6. Secondary Outcome: Change in Sleep Duration
Description: Data estimated using wrist actigraph.
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 37
hours | 1.11 (1.1)

7. Secondary Outcome: Change in SAFTEE Questionnaire Scores
Description: 128-item questionnaire asking participants to rank the level by which they have been bothered in the past week by common physical complaints people have, such as headaches, eye irritation, nasal congestion, etc. Items ranked on 5-point Likert scale ranging from 1 (not at all) to 5 (extremely). The total score is the average score of each item and ranges from 1-5; lower scores indicate less physical complaints. The change score is calculated as the change in scores between baseline and Week 15; the change score may range anywhere from 0-5.
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
score on a scale | 0.09 (0.17)

8. Secondary Outcome: Change in Physical Activity
Description: Estimated using accelerometer (count of steps).
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: Step Counts
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
Step Counts | -3576.17 (16,620.33)

9. Secondary Outcome: Change in Index of Self-Regulation (Sleep) Score
Description: 9-item questionnaire assessing self-regulation as it pertains to sleep. Items rated on 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). The total score is the average score for each item; higher scores indicate greater self-regulation.
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 41
score on a scale | -0.16 (0.61)

10. Secondary Outcome: Change in PROMIS Fatigue 6a Morning Score
Description: 6-item assessment of fatigue in the morning. Lowest score - 6; Highest score - 30; Lower score indicates less fatigue in the morning.
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 37
score on a scale | 4.95 (5.3)

11. Secondary Outcome: Change in PROMIS Fatigue 6a Evening Score
Description: 6-item assessment of fatigue in the Evening. Lowest score - 6; Highest score - 30; Lower score indicates less fatigue in the evening.
Time Frame: Baseline, Week 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Sleep Patients
Number analyzed (Participants) | 37
score on a scale | 5.36 (5.3)

ADVERSE EVENTS:
Time Frame: 15 Weeks
Description: A systematic method was used for determining adverese events using a standrad questionnaire in the REDCAp databse (C-DASH). Participants were queried for adverse events weekly at the end of their intervention session.
Arm/Group | Short Sleep Patients
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 4/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short Sleep Patients (N=44)
Minor skin irritation on wrist while wearing the accelerometer. (General disorders) | 2
Finger Injury (General disorders) | 1
Hospitalized for C-diff (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03596983/Prot_SAP_000.pdf